CLINICAL TRIAL: NCT03534674
Title: Validating a Vitamin D3 Supplementation Regimen Among Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Vitamin D3 Supplementation for AlloHSCT-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Raewyn Broady, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-03264
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention group will receive a single oral loading dose of 100,000 IU vitamin D3 on the day of hospital admission for aHSCT, with subsequent vitamin D3 2000 IU daily.
  Interventions: Dietary Supplement: vitamin D3
- Control (No Intervention): Participants assigned to the control group will be advised to take our current vitamin D regimen (2000 IU vitamin D3 daily).

INTERVENTIONS:
Dietary Supplement: vitamin D3 — a single oral loading dose of 100,000 IU vitamin D3 on the day of hospital admission for aHSCT, then 2000 IU vitamin D3 daily.
  Arms: Intervention

SUMMARY:
This study is to assess whether a single oral loading dose of 100,000 IU vitamin D3 prior to allogeneic hematopoietic stem cell transplant (aHSCT) can achieve optimal 25 hydroxy-vitamin D3(25-OH-D3) levels (>75nmol/L) at one month post aHSCT, and maintain adequate levels for at least three months, compared to our standard practice of 2000 IU vitamin D3 daily. 25-OH-D3 levels will be measured prior to vitamin D3 supplementation, and 30 as well as 100 days post vitamin D supplementation. We hypothesize that the intervention will prevent vitamin D insufficiency or deficiency in aHSCT recipients, therefore benefit aHSCT-associated morbidity, including osteoporosis.

DETAILED DESCRIPTION:
This is a randomized non-blinded single centre prospective clinical trial designed to validate whether a single oral loading dose of 100,000 IU vitamin D3 prior to allogeneic hematopoietic stem cell transplant (aHSCT) can achieve optimal 25 hydroxy-vitamin D3(25-OH-D3) levels (>75nmol/L) at one month post aHSCT, and maintain adequate levels for at least three months, compared to our standard practice of 2000 IU vitamin D3 daily.

84 patients will be enrolled. Following completion of all baseline data collection, participants will be randomized 1:1 to the intervention group or the control group on the admission day for aHSCT

Patients in the intervention group will receive a single oral loading dose of 100,000 IU vitamin D3, with subsequent vitamin D3 2000 IU daily. Patients assigned to the control group will receive our current standard of care, 2000 IU vitamin D3 daily.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing allogeneic stem cell transplantation at the Leukemia/BMT Program of British Columbia.
2. Age greater than or equal to 18 years.
3. Able to provide written informed consent.

Exclusion Criteria:

1. Hypercalcemia, hypervitaminosis D, or allergic/ sensitive to vitamin D.
2. Not meeting eligibility criteria to proceed with allogeneic stem cell transplantation as per the Leukemia/BMT Program of BC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of 100,000 IU vitamin D3 prior to aHSCT | 1 year
  To assess the efficacy (the proportion of patients achieving sufficient serum 25-OH-D3 level) after a single oral loading dose of 100,000 IU vitamin D3 prior to aHSCT, with subsequent vitamin D3 2000 IU daily, in preventing vitamin D insufficiency/deficiency in the first 100 days post-aHSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Raewyn Broady, MBChB, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided